CLINICAL TRIAL: NCT01545817
Title: Continuous Access to Advanced and Metastatic Renal Cell Carcinoma Therapy With Everolimus Post Pazopanib Treatment
Brief Title: Everolimus Post Pazopanib Treatment in Metastatic or Advanced Renal Cell Carcinoma
Acronym: CATChEz
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: As the therapeutic landscape in renal cell carcinoma is changing, it has become apparent that information gained so far by CATChEz study is sufficient.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 114907
Record Dates: First submitted 2011-11-17; First posted 2012-03-07 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal cell carcinoma (RCC), GW786034, Everolimus, Pazopanib, renal cancer, cancer, kidney cancer, hypernephroma, Grawitz tumor, renal adenocarcinoma.
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pazopanib followed by everolimus (Experimental): First line pazopanib, followed by second line everolimus
  Interventions: Drug: Pazopanib followed by everolimus

INTERVENTIONS:
Drug: Pazopanib followed by everolimus — All patients received Pazopanib (800 mg once daily orally continuous dosing) until disease progression then second line everolimus (10 mg once daily orally continuous dosing)
  Other Names: Pazopanib 1st line followed by everolimus 2nd line

SUMMARY:
Study to determine the efficacy, safety and tolerability of first-line pazopanib followed by second-line everolimus in metastatic and advanced renal cell carcinoma.

Due to changes in the RCC treatment landscape, info gained is no longer clinically relevant to patients. Data collected is deemed sufficient to meet objective.

DETAILED DESCRIPTION:
A non-randomised, open label, single-arm phase II study to evaluate the efficacy and safety of 1st-line pazopanib followed by 2nd-line everolimus in patients with previously untreated advanced or metastatic renal cell carcinoma. Subjects received initial therapy with pazopanib followed, on progression, by 2nd-line therapy with everolimus. Study treatment - sequential treatment with pazopanib followed by everolimus - to continue until disease progression, unacceptable toxicity, withdrawal of consent, or death.

ELIGIBILITY:
Inclusion criteria:

* Age >=18 years
* Histologically confirmed RCC with a clear-cell component
* Locally advanced or metastatic RCC
* At least one measurable lesion per RECIST 1.1 criteria, as determined by Computer Tomography (CT) Scan or Magnetic Resonance Imaging (MRI)
* No systemic therapy for advanced or metastatic RCC prior to enrollment
* Karnofsky Performance Status (KPS) ≥70
* Adequate baseline organ function
* A female was eligible to enter and participate in this study if she was of: non-childbearing potential, or negative serum pregnancy test with agreement to use adequate contraception during the study
* A male with female partner of childbearing potential must have vasectomy/agree to use effective contraception from 2 weeks prior to administration of the 1st dose of study treatment for a period of time after the last dose of study treatment
* Able to swallow and retain orally administered medication and must not have clinically significant GI abnormalities that may alter absorption

Additional inclusion criteria for starting everolimus:

* Disease progression must be within 6 months after stopping pazopanib
* At least one measurable lesion at the start of everolimus pe r RECIST 1.1 criteria, as determined by CT or MRI
* In case of central nervous system (CNS) progression or metastasis during pazopanib treatment: asymptomatic or neurologically stable, no requirement of steroids to control CNS symptoms, and no requirement of enzyme-inducing anticonvulsants within 4 weeks prior to the start of everolimus

Exclusion Criteria:

* Lactating female
* History of another malignancy (exception: patients disease-free for ≥3 years and patients with completely resected non-melanoma skin cancer or successfully treated in situ carcinoma)
* Symptomatic CNS metastases at baseline
* Clinically significant gastrointestinal abnormalities
* Moderate to severe hepatic impairment (Child Pugh Class C)
* Receiving chronic treatment with corticosteroids/other immunosuppressive agents
* Active bleeding, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin)
* Corrected QT interval (QTc) >480 msec using Bazett's formula
* Presence of any severe or uncontrolled medical conditions/infection
* Poorly controlled hypertension (defined as systolic blood pressure of >=140mmHg or diastolic blood pressure of >=90mmHg)
* History of cardiovascular disorders within the last 12 months (e.g. myocardial infraction or unstable angina), history of cerebrovascular events or pulmonary embolism within the last 6 months
* Active bleeding or bleeding susceptibility
* Known endobronchial lesion and/or lesions infiltrating major pulmonary vessels that increased the risk of pulmonary hemorrhage

Additional criteria for exclusion from the second-line everolimus treatment period:

- The subject felt by the investigator to be unsuitable (on the basis of health, compliance, or for any other reason) for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-04-19 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Australia (11):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Elizabeth Vale, South Australia
  - Novartis Investigative Site, Kurralta Park, South Australia
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Footscay, Victoria
  - Novartis Investigative Site, Frankston, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
- South Korea (2):
  - Novartis Investigative Site, Gyeonggi-do
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 patients were enrolled, all started first-line pazopanib treatment. Of these, 51 discontinued pazopanib and 38 continued to second-line everolimus treatment
Groups:
- Pazopanib: All patients were assigned to first-line treatment with pazopanib once daily. Pazopanib was supplied as 200 mg and 400 mg tablets. Pazopanib was administered once daily at the approved recommended dose of 800 mg/day (two 400 mg tablets, treatment taken once daily). The 200 mg tablets were provided to patients who needed dose adjustment.
- Everolimus: Patients who progressed during or within 6 months after stopping pazopanib treatment were eligible to then receive everolimus once daily (10 mg) as second-line treatment. Everolimus was supplied to the study sites as 5 mg and 10 mg tablets. The 5 mg tablets were provided to patients who needed dose adjustments.
Period: Pazopanib
Arm/Group | Pazopanib | Everolimus
Started | 74 | 0
Completed | 0 | 0
Not Completed | 74 | 0
Not completed — Disease progression | 51 | 0
Not completed — Adverse Event | 19 | 0
Not completed — Other reason | 4 | 0
Period: Everolimus
Arm/Group | Pazopanib | Everolimus
Started | 0 | 38
Completed | 0 | 0
Not Completed | 0 | 38
Not completed — Other reason | 0 | 7
Not completed — Disease progression | 0 | 25
Not completed — Adverse Event | 0 | 6

BASELINE CHARACTERISTICS:
Population: All Treated Subjects (ATS) population included all patients who received at least one dose of pazopanib.
Groups:
- All Patients: All patients were assigned to first-line treatment with pazopanib once daily. Patients who progressed during or within 6 months after stopping pazopanib treatment were eligible to then receive everolimus once daily as second-line treatment.
Arm/Group | All Patients
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) for the Everolimus Treatment Period Using RECIST
Description: Time between the date of first everolimus dose and date of disease progression or death (whichever comes first) in patients treated initially with pazopanib.
  Disease progression is measured by RECIST (Response Evaluation Criteria in Solid Tumors), which is at least a 20% increase in the sum of the target lesion longest diameters (LDs).
Time Frame: Throughout the study period, up to 4 years
Population: Intent to treat (ITT) population included all patients who received at least one dose of pazopanib and at least one dose of everolimus.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 38
months | 5.1 [3.4 to 6.8]

2. Secondary Outcome: Progression Free Survival (PFS) Rates
Description: PFS rates 3 and 6 months after date of first dose of second-line everolimus treatment.
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Survival probability
Arm/Group | All Patients
Number analyzed (Participants) | 38
Survival probability
  3 months | 0.737 [0.554 to 0.854]
  6 months | 0.355 [0.196 to 0.517]

3. Secondary Outcome: Objective Response Rate (ORR) for the Everolimus Treatment Period Using RECIST
Description: Percentage of patients with Complete or Partial Response at any time following the start of second-line everolimus treatment as per RECIST.
  RECIST Complete Response is defined to be a disappearance of all target lesion(s). RECIST Partial Response is defined to be at least a 30% decrease in the sum of the target lesion LDs.
Time Frame: Throughout the study, up to 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of Participants
Arm/Group | All Patients
Number analyzed (Participants) | 38
Percentages of Participants
  Complete response | 0.0 [0.00 to 9.3]
  Partial response | 7.9 [1.7 to 21.4]

4. Secondary Outcome: Objective Response Rate (ORR) for the Pazopanib Treatment Period Using RECIST
Description: Percentage of patients with Complete or Partial Response at any time following the start of first-line pazopanib treatment.
  RECIST Complete Response is defined to be a disappearance of all target lesion(s). RECIST Partial Response is defined to be at least a 30% decrease in the sum of the target lesion LDs.
Time Frame: Throughout the study period, up to 4 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Arm/Group | All Patients
Number analyzed (Participants) | 74
Percentages of participants
  Complete response | 6.8 [2.2 to 15.1]
  Partial response | 39.2 [28.0 to 51.2]

5. Secondary Outcome: Overall Survival of Everolimus (OSE)
Description: Time from first everolimus dose until death due to any cause
Time Frame: Throughout the study period, up to 4 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 38
months | 15.6 [9.9 to 25.3]

6. Secondary Outcome: Overall Survival From the Start (OSS) of Study Treatment
Description: Time from first pazopanib dose until death due to any cause in patients who received at least one dose of pazopanib followed by everolimus
Time Frame: Throughout the study, up to 4 years
Population: ATS
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pazopanib: All patients were assigned to first-line treatment with pazopanib once daily.
Arm/Group | Pazopanib
Number analyzed (Participants) | 74
Months | 35.7 [26.7 to NA] — not reached due to insufficient number of participants with events

7. Secondary Outcome: PFS for the Pazopanib Treatment Period Using RECIST
Description: Time from first pazopanib dose until disease progression or death from any cause (whichever occurred earlier), provided this occurred prior to the start of everolimus and within 6 months of last dose of pazopanib
Time Frame: Throughout the study period, up to 4 years
Population: ATS
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib
Number analyzed (Participants) | 74
Months | 11.0 [7.2 to 14.8]

ADVERSE EVENTS:
Time Frame: Adverse events for each intervention were assessed from the time of first dose of treatment to approximately one month after discontinuation of the last dose of treatment, up to 4 years.
Arm/Group | Pazopanib | Everolimus
All-Cause Mortality (participants affected / at risk) | 5/74 | 3/38
Serious Adverse Events (participants affected / at risk) | 47/74 | 16/38
Other Adverse Events (participants affected / at risk) | 73/74 | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=74) | Everolimus (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Incarcerated Hernia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 2
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Liver Injury (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Abscess Neck (Infections and infestations) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Pancreas Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4
Pulmonary Sepsis (Infections and infestations) | 0 | 1
Rectal Abscess (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 6 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Liver Function Test Abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vagus Nerve Paralysis (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=74) | Everolimus (N=38)
Anaemia (Blood and lymphatic system disorders) | 3 | 9
Palpitations (Cardiac disorders) | 4 | 1
Hypothyroidism (Endocrine disorders) | 8 | 0
Abdominal Pain (Gastrointestinal disorders) | 15 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 45 | 1
Dry Mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 14 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 9 | 1
Mouth Ulceration (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 37 | 6
Stomatitis (Gastrointestinal disorders) | 4 | 7
Vomiting (Gastrointestinal disorders) | 17 | 5
Asthenia (General disorders) | 1 | 2
Chest Pain (General disorders) | 1 | 2
Fatigue (General disorders) | 44 | 4
Gait Disturbance (General disorders) | 1 | 3
Influenza Like Illness (General disorders) | 4 | 1
Mucosal Inflammation (General disorders) | 8 | 6
Oedema Peripheral (General disorders) | 7 | 7
Peripheral Swelling (General disorders) | 5 | 1
Pyrexia (General disorders) | 7 | 3
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 0
Oral Candidiasis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 1
Urinary Tract Infection (Infections and infestations) | 9 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 3
Alanine Aminotransferase Increased (Investigations) | 6 | 0
Aspartate Aminotransferase Increased (Investigations) | 5 | 0
Blood Creatinine Increased (Investigations) | 2 | 2
Weight Decreased (Investigations) | 12 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 20 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophagia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 8 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7 | 2
Balance Disorder (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 5 | 1
Dysgeusia (Nervous system disorders) | 18 | 2
Headache (Nervous system disorders) | 13 | 3
Lethargy (Nervous system disorders) | 4 | 1
Presyncope (Nervous system disorders) | 4 | 0
Tremor (Nervous system disorders) | 5 | 0
Agitation (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 1
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 17 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 10 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 14 | 8
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 5 | 2
Hypertension (Vascular disorders) | 24 | 0
Hypotension (Vascular disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
the trial terminated early because the information gained from this study was sufficient to meet the objectives for which the study had been set up and would be no longer clinically relevant for the second-line management of RCC patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.